CLINICAL TRIAL: NCT06759155
Title: Phase II Clinical Trial of De-Intensified Therapy in Human Papilloma Virus (HPV) Associated Oropharyngeal Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, Mirabelle Sajisevi, Associate Professor, Division of Otolaryngology - Head & Neck Surgery, University of Vermont Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003257/UVMCC2405
Record Dates: First submitted 2024-12-19; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-11

CONDITIONS: OPSCC; Oropharyngeal Squamous Cell Carcinoma (SCC); HPV Associated Cancers
Keywords: radiation; de-intensify
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: Patients will be stratified into 4 groups depending on their risk factors. Groups A and be will not receive radiation (de-intensified), group C will receive a de-intensified level of radiation, group D will receive standard of care radiation (not de-intensified).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Very Low Risk (No Intervention): Patients with T1-T2 tumors which exhibit no adverse histological features (must have all of the following: negative margins, no perineural invasion or vascular invasion, 1 or fewer lymph nodes with metastasis ≤3 cm in size, negative for extranodal extension). Patients in this group will not receive any adjuvant treatment per standard of care.
- Low Risk (Experimental): Patients with T1-T2 tumors which exhibit no adverse histological features (must have all of the following: negative margins, no perineural invasion or vascular invasion), 2 lymph nodes with metastasis and/or lymph node metastasis 3.1-4cm in size, negative for extranodal extension, not "positive" or "intermediate" HPV ctDNA post-surgery. Patients in this group will not receive any adjuvant treatment. This is a de-intensified treatment, since NCCN guidelines recommend adjuvant radiation 60Gy for patients with a nodal metastasis greater than 3 cm in size or if there are multiple positive nodes
  Interventions: Radiation: de-intensified radiation
- Intermediate Risk (Experimental): Patients with any of the following - T3 tumors or T1-T2 tumors with additional risk factors (perineural invasion or vascular invasion), lymph node involvement greater than 4cm in size or with minimal extranodal extension (1-2mm), 3 or more lymph nodes with metastasis, "intermediate" or "positive" HPVctDNA post-surgery. Patients in this group will receive adjuvant radiation therapy at a de-intensified dose of 50Gy (as opposed to standard dose of 60Gy).
  Interventions: Radiation: de-intensified radiation
- High Risk (Experimental): Patients with tumors of any T or any N stage, which exhibit grossly positive margins or extensive extranodal extension. Patients in this group will receive standard of care treatment (per physician discretion, usually involves chemoradiation). Treatment for this group is not part of the protocol. Patient can elect to enroll on the imaging/HPV ctDNA surveillance component of the trial. Since this is not a de-intensified regimen, every effort will be made to reduce the number of patients in the high-risk category through careful baseline clinical exam and evaluation of imaging. In patients whom there is a concern for gross extranodal extension or that surgery will result in a grossly positive margin, they will be recommended to undergo a non-surgical route in order to avoid triple modality therapy.
  Interventions: Radiation: de-intensified radiation

INTERVENTIONS:
Radiation: de-intensified radiation — Adjuvant radiation will be administered on a de-intensified schedule.
  Arms: High Risk; Intermediate Risk; Low Risk

SUMMARY:
HPV-associated Oropharyngeal Squamous Cell Carcinoma (OPSCC) is a type of cancer that affects parts of the throat, like the tonsils and the base of the tongue. The treatments for OPSCC, which may include surgery, radiation, and chemotherapy, often cause serious side effects, such as loss of taste, dry mouth, and long-term problems with swallowing. These side effects can lower patients' quality of life and make it difficult for them to eat and speak normally.

This study aims to explore whether using lower doses of radiation after surgery can help improve long-term swallowing function in patients with HPV-positive OPSCC. By doing this, the study team hopes to reduce treatment-related side effects while maintaining good cancer control.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed or suspected HPV associated squamous cell carcinoma of the oropharynx.
* p16 immunohistochemistry is the surrogate marker for HPV positivity and will be scored as positive if there is strong and diffuse nuclear and cytoplasmic staining present in greater than 70% of the tumor specimen. (A negative result excludes the patient from the trial)
* In the case of equivocal p16, High Risk HPV (HR HPV), In-Situ Hybridization (ISH) / Polymerase Chain Reaction (PCR) may be performed to determine HPV positivity
* AJCC TNM 7th edition stage T1-T3, N0-N2b (or AJCC TNM 8th edition stage T1-T3 N0-N1) disease.
* Staging will be based on cross sectional imaging investigations and clinical exam.
* Patients who initially have an unknown primary but subsequently have a primary site identified on pathology after surgical resection may be included in the study.
* Multidisciplinary team decision to treat with primary transoral resection and neck dissection.
* Patients considered fit for surgery and adjuvant therapy.
* Aged 18 or over.
* Written informed consent provided.

Exclusion Criteria:

* HPV negative squamous cell carcinomas of the head and neck
* T4 and/or T1-T3 tumors where transoral surgery is considered not feasible or there is a high likelihood of positive margins.
* AJCC TNM 7th edition N2c-N3 nodal disease (or AJCC TNM 8th edition N2-N3 nodal disease) or high likelihood of gross extranodal extension.
* Patients for whom transoral surgery and neck dissection is not considered the primary treatment modality.
* Distant metastatic disease as determined by routine pre-operative staging radiological investigations e.g. CT thorax and upper abdomen or PET CT.
* Women who are pregnant or breastfeeding
* Prior history of radiation to head and neck

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Assess oncologic outcomes of a de-intensified post-surgical adjuvant treatment by measuring overall survival. | from enrollment to 5 year follow-up
  Overall survival will be monitored.
Safety and tolerability | from enrollment to 5 year follow-up
  The study will use the CTCAE version 5.0 for reporting of non-hematologic adverse events.
Assess oncologic outcomes of a de-intensified post-surgical adjuvant treatment by measuring progression free survival. | from enrollment to 5 year follow-up
  Assess oncologic outcomes of a de-intensified post-surgical adjuvant treatment by measuring progression free survival.
Assess oncologic outcomes of a de-intensified post-surgical adjuvant treatment by measuring locoregional control. | from enrollment to 5 year follow-up
  Locoregional control (LRC) is defined as time from treatment initiation to local or regional recurrence

SECONDARY OUTCOMES:
Evaluate how changes in serum HPV ctDNA are associated\ with HPV-positive OPSCC recurrence | from enrollment to 5 year follow-up
  ctDNA will be measured at baseline and at several points during follow-up. The sensitivity, specificity and concordance of the HPV ctDNA results in relation to the clinical and pathologic disease status (presence/absence) will be corelated.

IPD SHARING:
Plan to Share IPD: Undecided